CLINICAL TRIAL: NCT06585943
Title: The I-Score (Intensive Stroke Cycling for Optimal Recovery and Economic Value) Trial
Brief Title: I-Score: Intensive Stroke Cycling for Optimal Recovery and Economic Value
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Susan Linder, Associate Professor, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 23-1262
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Stroke
Keywords: aerobic exercise; physical therapy; occupational therapy
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: prospective, single-center, parallel group, rater-blind, pragmatic randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Forced Rate Exercise + Rehabilitation (Active Comparator): The forced rate exercise+rehab group (N=33) will complete FE on the cycle designed to augment pedaling rate to >75 revolutions per minute (RPM). Target heart rate zone will be set to 60-80% of heart rate (HR) reserve. The session will consist of a 5-min warm-up, 35-min main exercise set, and 5-min cool down. Following FE, abbreviated sessions of motor learning-based training will be administered by a neurologic OT and PT experienced in stroke rehabilitation, with 30 min focused on restoration of UE function (OT) and 15 min focused on LE motor function/ gait training (PT).
  Interventions: Behavioral: Forced Rate Exercise + Rehab
- Rehabilitation (Active Comparator): The rehab group will receive consecutive, full-length sessions of motor learning-based training, administered by a neurologic OT and PT experienced in stroke rehabilitation, with 45 min focused on restoration of UE function (OT) and 45 min focused on LE motor function/ gait training (PT).
  Interventions: Behavioral: Rehabilitation

INTERVENTIONS:
Behavioral: Forced Rate Exercise + Rehab — The FE+rehab group (N=33) will complete FE on the cycle designed to augment pedaling rate to >75 RPM. Target heart rate zone will be set to 60-80% of HR reserve. The session will consist of a 5-min warm-up, 35-min main exercise set, and 5-min cool down. Following FE, abbreviated sessions of motor learning-based training will be administered by a neurologic OT and PT experienced in stroke rehabilitation, with 30 min focused on restoration of UE function (OT) and 15 min focused on LE motor function/ gait training (PT).
  Arms: Forced Rate Exercise + Rehabilitation
Behavioral: Rehabilitation — The rehab group will receive consecutive, full-length sessions of motor learning-based training, administered by a neurologic OT and PT experienced in stroke rehabilitation, with 45 min focused on restoration of UE function (OT) and 45 min focused on LE motor function/ gait training (PT).
  Arms: Rehabilitation

SUMMARY:
Traditional rehabilitation approaches are time and personnel intensive and costly, and leave ~75% of stroke survivors with residual disability. We propose a clinical trial to determine effects of forced aerobic exercise (FE; i.e., mechanically supplemented) in facilitating upper and lower extremity motor recovery post-stroke in an outpatient rehabilitation setting, to elucidate neural and biochemical substrates of FE-induced motor recovery, and to evaluate cost effectiveness of a FE-centered intervention compared to traditional stroke rehabilitation. The global effect of FE has the potential to enhance recovery in a growing population of stroke survivors in a cost-effective manner, thus accelerating its clinical acceptance.

DETAILED DESCRIPTION:
Traditional rehabilitation approaches following stroke involve 1:1 motor learning-based training to facilitate recovery of upper extremity (UE) and lower extremity (LE) function. These time- and personnel-intensive approaches are costly, yet leave ~75% of stroke survivors with residual disability. More effective alternative approaches to facilitate motor recovery following stroke have not been adopted clinically due to excessive time and cost. To advance clinical care, both effectiveness and cost of a candidate intervention must be considered simultaneously. Aerobic exercise (AE) is known to improve cardiovascular function following stroke and central nervous system (CNS) function in older adults and neurological populations. Strong theoretical arguments suggest that AE may facilitate motor recovery following stroke. A protocol that rigorously tests this theory in the subacute stroke population is warranted. Animal studies, coupled with our preliminary data, indicate a specific type of exercise - forced aerobic exercise (FE), where volitional movements are mechanically supplemented - improves motor recovery following stroke. The mechanical assistance provided by FE enables patients to achieve a more rapid and consistent exercise pattern beyond their volitional capabilities while maintaining their aerobic effort within a beneficial range. In our initial studies, persons completing FE cycling followed by a reduced dose of UE motor task practice exhibited greater recovery of UE motor function compared to those completing unassisted AE and motor task practice or extended sessions of motor task practice alone. Animal studies have shown that FE triggers the release of brain-derived neurotrophic factor (BDNF) and insulin-like growth factor-1 (IGF-1), thought to be critical building blocks for neuroplasticity. Project Hypothesis: FE facilitates high-intensity AE, which triggers growth factors essential for neuroplasticity, thereby 'priming' the CNS to facilitate motor recovery associated with motor retraining therapies. We propose a prospective, pragmatic clinical trial to determine effects of FE in facilitating UE and LE motor recovery post-stroke in an outpatient rehabilitation setting, to elucidate neural and biochemical substrates of FE-induced motor recovery, and to evaluate cost effectiveness of a FE-centered intervention compared to traditional stroke rehabilitation.

Aim 1: Determine effects of FE+rehab vs. time-matched rehab on the recovery of UE motor function.

Aim 2: Determine effects of FE+rehab vs. time-matched rehab on recovery of lower extremity motor function.

Aim 3: Determine effects of FE+rehab vs. rehab on electrophysiological and biochemical markers of neuroplasticity.

Aim 4: Evaluate cost-effectiveness of FE+rehab vs. rehab. The global effect of FE has the potential to enhance recovery in a growing population of stroke survivors in a cost-effective manner, thus accelerating its clinical acceptance. Our mechanistic aim will elucidate the effects of each approach on substrates underlying neuroplasticity.

ELIGIBILITY:
Sixty-six individuals with chronic stroke able to provide informed consent who meet the following criteria for inclusion will be recruited from the Cleveland Clinic:

1. 3-9 months following single ischemic or hemorrhagic stroke confirmed with neuroimaging (ie: first-time stroke)
2. Fugl-Meyer motor score 19-55 in the involved UE
3. Fugl-Meyer score <34 in the involved LE demonstrating residual hemiparesis
4. Ambulatory ≥ 20 meters with no more than contact guard assistance
5. 18-85 years of age

Exclusion criteria include:

1. hospitalization for myocardial infarction, heart failure or heart surgery within 3 months
2. cardiac arrhythmia
3. hypertrophic cardiomyopathy
4. history of multiple strokes
5. actively undergoing physical or occupational therapy or enrolled in another interventional study
6. severe aortic stenosis
7. untreated deep vein thrombosis or pulmonary embolus
8. unstable angina
9. uncontrolled hypertension
10. implanted pacemaker or defibrillator
11. dyspnea at rest
12. clinically significant neurologic condition/diagnosis other than stroke
13. recent history of elicit drug or alcohol misuse or significant mental health illness
14. significant contractures
15. anti-spasticity injection within 3 months of enrollment
16. skull hardware (e.g. screws/plates) or prior craniotomies that could shunt current flow altering EEG measures
17. other contraindication to exercise or EEGs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Upper Extremity Fugl-Meyer Motor Assessment | Baseline to end of treatment at 12 weeks and end of treatment + 6 months
  Impairment-based measure of the upper extremity post-stroke.
Gait Velocity | Baseline to end of treatment at 12 weeks and end of treatment + 6 months
  Gait velocity obtained using motion capture.
Plasma IGF-1 | Before and after first and 24th treatment session
  Blood biomarker for neuroplasticity
Serum BDNF | Before and after first and 24th treatment session
  Blood biomarker for neuroplasticity
electroencephalograms | Baseline and end of treatment at 12 weeks
  Electroencephalograms will be obtained to determine the degree of active engagement of different cortical areas during active/passive UE and LE movements
electroencephalograms | Baseline and end of treatment at 12 weeks
  Electroencephalograms will be obtained to determine the degree of active engagement of different cortical areas under each cycling condition
electroencephalograms | Baseline and end of treatment at 12 weeks
  Electroencephalograms will be obtained to quantify inter-area communication and direction of information flow.
Incremental cost-effectiveness ratio | baseline to end of treatment at 12 weeks and baseline to end of treatment + 6 months
  Incremental cost-effectiveness ratio (ICER) expressed as cost per quality of life years (QALY) will be computed using a healthcare perspective.
Stroke Impact Scale | Baseline to end of treatment at 12 weeks and end of treatment + 6 months
  Self-reported quality of life measure, normalized to a score from 0-100 with higher scores indicative of better self-reported quality of life

SECONDARY OUTCOMES:
Action Research Arm Test | Baseline to end of treatment at 12 weeks and end of treatment + 6 months
  Measure of upper extremity gross and fine motor function post-stroke
Biomechanical Dexterity Task | Baseline to end of treatment at 12 weeks and end of treatment + 6 months
  Force tracking task - accuracy within targeted range
Biomechanical measure of maximum grasp force | Baseline to end of treatment at 12 weeks and end of treatment + 6 months
  maximum grasp force measured with force transducer
Bimanual Dexterity Task | Baseline to end of treatment at 12 weeks and end of treatment + 6 months
  Time to complete task when separating 2 force transducers
Six minute walk test | Baseline to end of treatment at 12 weeks and end of treatment + 6 months
  Measure of walking capacity
Lower Extremity Fugl-Meyer Motor Assessment | Baseline to end of treatment at 12 weeks and end of treatment + 6 months
  Impairment-based measure of the lower extremity post-stroke.
Biomechanical Gait Analysis | Baseline, end of treatment at 12 weeks, end of treatment + 6 months
  Biomechanical assessment of the following spatio-temporal components of gait using motion capture: % of gait cycle spent in swing and stance phases, and in single and double limb support.
Biomechanical Gait Analysis | Baseline, end of treatment at 12 weeks, end of treatment + 6 months
  Biomechanical assessment of gait cadence (steps/minute)
Biomechanical Gait Analysis | Baseline, end of treatment at 12 weeks, end of treatment + 6 months
  Biomechanical assessment of stride length
Biomechanical Gait Analysis | Baseline, end of treatment at 12 weeks, end of treatment + 6 months
  Biomechanical assessment of the following components of gait kinetics using motion capture: 1) peak anterior-posterior propulsion forces, 2) peak anterior-posterior braking forces, 3) peak vertical ground reaction forces, 4) peak lateral ground reaction forces.
Biomechanical Gait Analysis | Baseline, end of treatment at 12 weeks, end of treatment + 6 months
  Biomechanical assessment of the following components of gait kinetics using motion capture: 1) total hip extension moment 2) total knee extension moment, 3) total ankle plantarflexion extension moment
Biomechanical Gait Analysis | Baseline, end of treatment at 12 weeks, end of treatment + 6 months
  Biomechanical assessment of the following components of gait kinetics during stance phase using motion capture: 1) total hip extension power 2) total knee extension power, 3) total ankle plantarflexion extension power
Biomechanical Gait Analysis | Baseline, end of treatment at 12 weeks, end of treatment + 6 months
  Biomechanical assessment of the following kinematic components of gait using motion capture: hip flexion/extension, knee flexion/extension, ankle plantar- and dorsi-flexion
Plasma BDNF | Before and after first and 24th session
  Blood biomarker for neuroplasticity
Somatosensory evoked potentials | Baseline
  lower extremity somatosensory evoked potentials
Modified Rankin Scale | Baseline to end of treatment at 12 weeks and end of treatment + 6 months
  Measure of disability
Peak oxygen consumption (Peak VO2) | Baseline to end of treatment at 12 weeks
  Measure of cardiorespiratory function
Patient-Reported Outcomes Measurement Information System (PROMIS) Computerized Adaptive Test (CAT) v 2.0 Physical Function | Baseline to end of treatment at 12 weeks and end of treatment + 6 months
  Self-reported quality of life measure of physical function computed as normalized T-scores (1-100 range), with higher scores indicative of greater self-reported quality of life
Patient-Reported Outcomes Measurement Information System (PROMIS) Computerized Adaptive Test (CAT) v 2.0 Ability to Participate in Social Roles | Baseline to end of treatment at 12 weeks and end of treatment + 6 months
  Self-reported quality of life measure computed as a normalized T-score (0-100 range), with higher scores indicative of greater self-reported participation

CONTACTS AND LOCATIONS:
Overall Officials: Susan Linder, PT, DPT, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No